CLINICAL TRIAL: NCT02377453
Title: A Longitudinal Study of Function and Participation in Patients With Stroke: An Integrated Brain Imaging and Biomechanical Analysis
Brief Title: A Longitudinal Study of Function and Participation in Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-5783B
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: stroke; participation; brain imaging; biomechanical
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Control: Healthy adult
- Experimental: Experimental: patients with stroke

SUMMARY:
A longitudinal study of function and participation in patients with stroke: An integrated brain imaging and biomechanical analysis

DETAILED DESCRIPTION:
Brain damage may lead to various motor deficits, which further influence the function and participation. Cerebral vascular accident (CVA) is the common disorder for acquired brain damage. Neural network in patients with brain damage could also be used to determine their clinical behavior by identifying altered neural network associated with behavioral improvement. The investigators hypothesize that the level of brain image and biomechanical will change with time in patients with stroke. Under this hypothesis, the measures of biomechanical change are correlated with neural changes. The aim of this study is to investigate the function and participation in patients with stroke evaluated by clinical measures, biomechanical, psychological, physiological and multimodal brain image. The primary goal of this study is to establish, evaluate and follow-up biomechanical- and image-based biomarkers for the impairment of function and participation information processing present in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stroke
2. Aged 20-80 years old
3. Both ischemic stroke and hemorrhage

Exclusion Criteria:

1. Contraindication to MRI, such as metallic implant
2. History of psychiatric disease
3. Received Botulinum toxin (BTX-A) injection or surgery in recent six months
4. Severe psychological impairments, such as mental retardation or severe Communication problems
5. Progressive disorders, such as neurodegenerative disease
6. Active medical disease, such as infection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control and experimental groups
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of biomechanical measurement for Healthy adult and patients with stroke in 6 months and 12 months | baseline, 6 months, 12 months
  Muscle tone, Muscle strength and Kinematic analysis for upper limb and gait analysis

SECONDARY OUTCOMES:
Change from baseline of functional magnetic resonance imaging (fMRI) analysis in 6 months and 12 months | baseline, 6 months, 12 months
  fc(functional connectivity)MRI at resting, active-task fMRI. diffusion tensor imaging (DTI)
Change from baseline of psychological in 6 months and 12 months | baseline, 6 months, 12 months
  CANTAB touchscreen
Change from baseline of body composition in 6 months and 12 months | baseline, 6 months, 12 months
  InBody230 Body Composition Analyzer
Change from baseline of severity in 6 months and 12 months | baseline, 6 months, 12 months
  Brunnstrom stage classification, Modified Ashworth Scale and National Institute of Health Stroke Scale
Change from baseline of body in 6 months and 12 months | baseline, 6 months, 12 months
  Minimal Mental State Examination, Beck Depression Inventory-II, Fugl-Meyer assessment, Pediatric Berg Balance Scale, Action Research Arm Test and Box and Block Test
Change from baseline of activity in 6 months and 12 months | baseline, 6 months, 12 months
  Barthel Index, Wolf motor function test, Motor activity log, Walking test, Timed 'Up & Go' test and Functional Independence Measure
Change from baseline of participation in 6 months and 12 months | baseline, 6 months, 12 months
  Adaptive behavior assessment system and Nottingham Health Profile
Change from baseline of quality of life in 6 months and 12 months | baseline, 6 months, 12 months
  Stroke Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No